CLINICAL TRIAL: NCT04692337
Title: Ommaya Reservoir Placement for Brain Tumor Biomarker Access
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-009226; R33NS122096 (NIH); NCI-2021-02766 (Other: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2020-12-29; First posted 2020-12-31 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ommaya Reservoir placement (Experimental): Subjects undergoing surgery for a confirmed or suspected brain tumor will have an Ommaya Reservoir placed at the time of surgery.
  Interventions: Procedure: Intra-operative Ommaya Reservoir placement

INTERVENTIONS:
Procedure: Intra-operative Ommaya Reservoir placement — An Ommaya reservoir is a small device implanted under the scalp that enables percutaneous access to cerebrospinal fluid.

SUMMARY:
The purpose of this study is to determine the safety and feasibility of intra-operative Ommaya Reservoir placement during a clinically indicated operation for brain tumor. The Ommaya reservoir will facilitate a longitudinal access to cerebrospinal fluid (CSF) for analysis of potential biomarkers for brain tumor research and individualized monitoring.

DETAILED DESCRIPTION:
Most brain tumors remain incurable. Progress in clinical trials to identify better treatments has been slow. We hypothesize that longitudinal CSF access can provide insights regarding tumor identity, behavior and the efficacy of candidate therapies. Although multiple studies have evaluated CSF from patients with brain tumors, very few have collected CSF at multiple timepoints throughout the course of disease. However, multiple samples over time are needed to determine if candidate biomarkers accurately reflect the evolution of disease. CSF is typically obtained via lumbar puncture which is inconvenient and often uncomfortable. This protocol will evaluate the safety and feasibility of placing Ommaya reservoirs at the time of surgery. It is anticipated that reducing barriers to CSF access through placement of an Ommaya reservoir may expedite brain tumor research and facilitate the development of individualized treatment strategies.

An Ommaya Reservoir will be placed during a planned brain tumor operation. Following the routine portion of the planned procedure, the Ommaya reservoir will be placed under the scalp with the catheter tip placed either within the ventricle or the resection cavity. Presence of the Ommaya reservoir will enable CSF to be easily accessed at any time in the future. It is expected that CSF will be collected at 2 or more timepoints. CSF will be stored in the Mayo Clinic neuro-oncology biorepository and made available in a de-identified manner for multiple research projects. The patient and his/her provider(s) may take advantage of the Ommaya reservoir and/or banked CSF samples to facilitate participation in any relevant IRB-approved research study(s), and/or to facilitate individualized management. The details of each time the Ommaya is accessed will be documented as part of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Clinical and radiographic evidence suggesting a diagnosis of a brain tumor.
* Planned neurosurgical procedure resection of suspected or previously diagnosed brain tumor as part of routine clinical care.
* Willing to undergo neurosurgical resection at Mayo Clinic (Rochester, MN).
* Willingness of the patient or an authorized representative to provide informed consent
* Patient is willing to have their Ommaya sampled on at least 2 future occasions.
* Patients is willing to have CSF banked through the neuro-oncology biorepository (requires a separate signature)

Exclusion Criteria:

* Vulnerable populations including pregnant women, prisoners and individuals <18 years old.
* Patients who are not appropriate candidates for surgery due to current or past medical history or uncontrolled concurrent illness.
* Prior history of any wound infection
* Any patient who the surgeon feels is not an optimal candidate for Ommaya reservoir placement. Such reasons could (but need not necessarily) include factors related to surgical anatomy, clinical evidence of significant immunosuppression, and/or elevated risk of wound infection due to diabetes, smoking history, morbid obesity, or any other concerns.
* Any patient for whom a clinical contraindication exists to a lumbar puncture (LP) will be excluded from the LP portion of this protocol, but would still be eligible for an Ommaya reservoir if they meet the inclusion criteria of the study. For example, a patient with a large posterior fossa mass lesion at risk of herniation, or a patient with coagulopathy, or other contraindication to lumbar puncture would not be eligible to participate via use of lumbar puncture for CSF access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Collection of serial CSF samples for biobanking and biomarker discovery and validation - proportion of patients | Through study completion, approximately 42 days
  Assessed by the proportion of patients for whom longitudinal CSF can be collected.
Collection of serial CSF samples for biobanking and biomarker discovery and validation - number of times | Through study completion, approximately 42 days
  Assessed by the number of times longitudinal CSF collection occurred
Collection of serial CSF samples for biobanking and biomarker discovery and validation - volume obtained | Through study completion, approximately 42 days
  Assessed by the volumes obtained at each Ommaya tap.

SECONDARY OUTCOMES:
Incidence of Adverse Events of intra-operative Ommaya Reservoir placement | Through study completion, approximately 42 days
  Number of subjects to develop persistent adverse events deemed related (possibly, probably, definitely) to the insertion or use of Ommaya Reservoirs. Adverse events will be measured by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Scope of CSF biomarkers | Through study completion, approximately 42 days
  Assessed by the number of assays run for each patient and the number of times the assays successfully detected an analyte under consideration as a candidate biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Terry C. Burns, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Protocol details and individualized de-identified patient data will be provided as supplemental files in the resulting publication. Any additional information not otherwise provided may be requested from the primary investigator.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Any time after publication.
Access Criteria: Requests will be honored that could help advance the care of patients with brain tumors.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials